CLINICAL TRIAL: NCT02940938
Title: Study on Changes of Pulse Oximeter Plethysmographic Amplitude Induced by Respiration in Pediatric Patients: the Effect of Contacting Force
Brief Title: Study on Changes of Pulse Oximeter Plethysmographic Amplitude Induced by Respiration in Pediatric Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H1609-067-791
Record Dates: First submitted 2016-10-19; First posted 2016-10-21 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2016-12

CONDITIONS: Children Under General Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children under general anesthesia (Experimental): During general anesthesia without surgical stimuli, pulse oximeter sensor is applied with gradually increased contact force, from 0 to maximal 1.5N (increase by about 0.2N), at an index finger and POP waveform is obtained for 60 seconds at each contact force. Delta POP will be calculated and compared.
  Interventions: Other: Applying pulse oximeter sensor

INTERVENTIONS:
Other: Applying pulse oximeter sensor — During general anesthesia, pulse oximeter sensor is applied with gradually increased contact force, from 0 to 1.5N (increase by about 0.2N), at an index finger and POP waveform is obtained for 60 seconds.

SUMMARY:
The purpose of this study is to evaluate the variations of respiratory changes in pulse oximeter plethysmographic amplitude (delta POP) according to different contact forces between finger and sensor of pulse oximeter. During general anesthesia without surgical stimuli, pulse oximeter sensor is applied with serial contact force, from 0 to maximal 1.5N (increased by 0.2N) and POP waveform is obtained for 60 seconds. Delta POP will be calculated and compared.

ELIGIBILITY:
Inclusion Criteria:

* children who are aged between 2 and 5 years
* no cardiopulmonary and vascular diseases
* obtained written informed consent from their guardians
* no hemodynamic instability from massive bleeding

Exclusion Criteria:

* significant cardiopulmonary or vascular disease
* significant hemodynamic instability due to massive bleeding etc.
* cyanotic patients

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Respiratory changes in pulse oximeter plethysmographic amplitude measured | about 3 minutes after anesthetic induction without surgical stimuli
  Respiratory changes in pulse oximeter plethysmographic amplitude measured by pulse oximeter sensor with different contact force

SECONDARY OUTCOMES:
Amplitude of pulse oximeter plethysmography | about 3 minutes after anesthetic induction without surgical stimuli
  Amplitude of pulse oximeter plethysmography measured by pulse oximeter sensor with different contact force

CONTACTS AND LOCATIONS:
Locations (1):
- SNUH, Seoul, Jongro Gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided